CLINICAL TRIAL: NCT02332005
Title: Twelve-Month Chronic Efficacy and Safety of Diepalrestat in Adult Subjects With Diabetic Peripheral Neuropathy (DPN), A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: 12-Month Efficacy and Safety of Diepalrestat in Adults With Diabetic Peripheral Neuropathy, a DB, Placebo-Controlled Study
Acronym: DE-DPN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NeuromaxBionevia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NM-ARI-231
Record Dates: First submitted 2015-01-02; First posted 2015-01-06 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 150 mg (Active Comparator): 150 mg diepalrestat choline administered as twice daily dosing morning and evening with an oral tablet of either 150 mg diepalrestat choline or placebo
  Interventions: Drug: diepalrestat choline
- Group 2 300 mg (Active Comparator): 300 mg diepalrestat choline administered as twice daily dosing morning and evening with an oral tablet of 150 mg diepalrestat choline
  Interventions: Drug: diepalrestat choline
- Group 3 (Placebo Comparator): Tablet administered twice daily morning and evening containing placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: diepalrestat choline — aldose reductase inhibitor
  Other Names: BNV-222
  Arms: Group 1 150 mg; Group 2 300 mg
Drug: Placebo — Placebo
  Arms: Group 3

SUMMARY:
An interventional study to investigate the efficacy and safety of diepalrestat (BNV-222) in diabetic patients with diabetic peripheral neuropathy. Subjects will receive twice daily an oral dose of diepalrestat, an aldose reductase inhibitor, or placebo to investigate the effect on motor nerve conduction velocity (MNCV) and symptomatic clinical responses over 12 months of treatment. Subjects will be assessed at screening and baseline, with office visits every 12 weeks, for a total of 6 visits. The study will explore in a double-blind fashion, the effect of two doses of diepalrestat, 150 and 300 mg, to reduce the loss in nerve conduction velocity that is expected to be demonstrated in the group randomized to placebo treatment for up to 12 months.

DETAILED DESCRIPTION:
This 12 month double-blind, randomized, placebo-controlled, parallel group efficacy and safety study will enroll 400 adult diabetic subjects with diabetic peripheral neuropathy (DPN) to investigate the effect of diepalrestat (BNV-222) 150 mg, 300 mg, or placebo on MNCV and patients' perception of nerve function over 12 months as measured by VAS scales and composite clinical outcome patient reported scales that evaluate numbness, tingling, cramping, paresthesiae, hyperesthesia, coldness, weakness and spontaneous pain perception of upper and lower extremities, and the effects on other measures of nerve motor and sensory conduction. Subjects will be assessed at screening and baseline, with office visits every 12 weeks, for a total of 6 visits. Subjects will be assessed by testing motor nerve conduction velocity and other assessments at each office visit. A subgroup of 24 patients will be selected for pharmacokinetic (PK) testing for up to 48 hours with additional blood draws on Day 7 and 14. This study will investigate the ability of diepalrestat to reduce the ongoing deterioration of nerve function which is a hallmark of the DPN process.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or type 2 diabetes mellitus that is controlled by oral or parenteral hypoglycemic agents or diet.
* Patients with diabetes that is stable and controlled (HbA1C ≤ than 10 %) with no new symptoms associated with diabetes within previous 3 months.
* Patients diagnosed with neuropathy who have abnormalities in 2 of 3 categories (signs, symptoms, and objective tests of nerve conduction studies or quantitative sensory threshold testing).
* Patients on pain medication (prescribed analgesics), stable for at least 3 months before study entry or pain treatment naive.
* Patients with at least mild painful symptoms of diabetic neuropathy for at least 1 year duration, but not longer than 10 years duration.
* Able to withstand the fundus evaluation during ophthalmology testing

Exclusion Criteria:

* A condition that would preclude a patient for participation in the study in opinion of investigator, e.g., unstable medical status including glycemic control and blood pressure.
* Any neurological disorder that may confound assessment of diabetic peripheral neuropathy such as radiculopathies. multiple sclerosis, myelopathies.
* Ongoing severe peripheral arterial diseases, skin ulcers, or amputation in the lower extremities.
* Neuropathy findings due to any of the following: alcohol abuse, liver or renal disease, toxic exposure, endocrine, metabolic or nutritional disorders, inflammatory diseases, or monoclonal gammopathies.
* Patients with absent peroneal nerve response.
* Other pain that may confound assessment of neuropathic pain.
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
change from baseline in peroneal motor nerve conduction velocity | 12 months

SECONDARY OUTCOMES:
change from baseline in patient-reported Visual Acuity Scales | 12 months
  Patients' perception of pain, numbness, tingling, weakness of the foot, ataxia, upper limb symptoms and sensory symptoms assessed by pinprick, light touch, vibration, and temperature
change from baseline in patient-reported responses to Toronto Clinical Neuropathy Score (TCNS) | 12 months
  TCNS component measures of symptomatic changes in pain, numbness and other measures
change from baseline in quality of life administered by SF-36 instrument | 12 months
  patient global impression of quality of life assessed by the SF-36 short form
change from baseline in median conduction velocity measurements | 12 months
  conduction velocity measures including median MNCV,
change in visual acuity compared to baseline | 12 months
  Change in visual acuity over 12 months compared to baseline, change in diabetic retinopathy in the dilated eye
change from baseline in MFWL conduction velocity measurement | 12 months
  change from baseline in median F wave latency (MFWL)
change from baseline in VPT conduction velocity measurement | 12 months
  change from baseline in Vibration Perception Threshold (VPT)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Mockot, MD, Study Director — NeuroMax Ltd.
Locations (26):
- Russia (26):
  - City Hospital No 40 of the Kurortny District, Saint Petersburg, Sestroretsk
  - Northern State Medical University, Arkhangelsk
  - Health Services Severstal, Cherepovets
  - Kemerovo Regional Clinical Hospital, Kemerovo
  - Endocrinology Dispensary, Moscow
  - Morozovskaya Children City Hospital of Moscow, Moscow
  - I M Sechenov First Moscow State Medical University, Moscow
  - IM Sechenov First Moscow State Medical University, Moscow
  - City Clinical Hospital No 71, Moscow
  - Central Clinical Hospital No 1 of JSC Russian Railway, Moscow
  - City Clinical Hospital No 50, Moscow
  - The Federal Bureau of Medical and Social Expertise, Moscow
  - Perm State Medical Academy, Perm
  - VA Baranov Respublical Hospital, Petrozavodsk
  - Rostov State Medical University, Rostov-on-Don
  - Imc Sogaz, Saint Petersburg
  - Medical Center Reavita, Saint Petersburg
  - City Hospital of the Holy Martyr Elizabeth, Saint Petersburg
  - Nikolaev Hospital, Saint Petersburg
  - City Polyclinic No 20, Saratov
  - Bashkir State Medical University, Ufa
  - Central City Clinical Hospital, Ulyanovsk
  - State Medical University, Volgograd
  - Regional Clinical Hospital, Yaroslavl
  - NV Solovyov Clinical Emergency Hospital, Yaroslavl
  - Clinic of Neurology, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes